**Protocol Title:** SSRI Effects on Depression and Immunity in HIV/AIDS

NCT Number: NCT02620150

**Document:** Statistical Analysis Plan

**Document Date:** March 10, 2015

### C.3 Research Design and Methods

**Aim 1** Determine the effects of an SSRI on innate immunity and inflammation in depressed HIV seropositive individuals.

# C.3.1 Summary

This will be the first placebo-controlled RCT to determine the immunomodulatory effects of SSRI therapy among a contemporary, urban cohort of HIV-seropositive individuals whose viral load is well controlled, yet still experiences immune dysregulation due to co-morbid depression and HIV infection Comparing the two depressed groups that are randomly assigned to receive SSRI or placebo will allow us to address novel aims: can SSRI treatment and improvement of depression reverse the immune dysregulation of depression and HIV. Comprehensive biomarkers of innate immunity, and inflammation will be assayed via blood draw at baseline and at 2, 4, and 10 weeks. Additionally, we will monitor adherence to SSRI and antiretroviral medications in all participants using contemporary methodology (i.e., self-reported doses taken and missed, medication electronic monitoring system (MEMS) caps, and, for HIV, plasma viral load).

**Aim 1A.** Determine whether an SSRI upregulates innate immunity in depressed HIV seropositive individuals. <u>Hypothesis:</u> SSRI is superior to placebo in restoring biomarkers of innate immune suppression (LUNK and intracellular IFNy in NK cells).

Previously we demonstrated that major depression is associated with significant reductions in NK cell activity and resolution of depression resulted in improvement of LUNK (for details see C1.7, C1.8). SSRI enhances LUNK ex vivo (for details see C1.9.a). In addition as a part of our recent project (RO1 MH82670) we demonstrated that increase in severity of depression is associated with decrease in absolute numbers of total NK cells (p=0.008), reduction in perforin+ NK cells (p=0.009) and reduced expression of activation receptors NKP30+ (p=0.011) and NKP46+ (p=0.049) (unpublished observations). NK cell functions are also affected by HIV infection in several ways including decreased cytotoxic activity, changes in receptor expression and cytokine production (123-125). Although NK functions are partially restored by cART(44, 123), several studies demonstrated that recovery is incomplete. NK cells from HIV positive individuals with sustained viral suppression by cART do not completely recover in numbers (44), continue to have increased activation/degranulation profiles (46), show decreased receptor expression (NKp46 and NKp30) (126) and decreased cytokine production (IFNγ, TNF-α) (127).

In this aim we will assess NK cell functions in HIV positive individuals on stable cART at baseline and after 2, 4, and 10 weeks of SSRI therapy. NK cell function will be assessed by the standard chromium release assay, established in our laboratory, using K562 target cells and peripheral blood mononuclear cells (PBMC) at effector to target cell ratios of 6.25 - 50. Percent lysis values will be normalized for percent NK cells within the PBMC preparations and are expressed as lytic units (LU) per  $10^7$  NK cells or LUNK as previously described (41, 71, 72). In addition intracellular IFN $\gamma$  will be assessed as described (42) (also see letter from Dr. Luis J. Montaner) in stimulated PBMCs. The number of IFN $\gamma$ <sup>+</sup> NK cells will be assessed by flow cytometry gated on CD45<sup>+</sup>/CD3<sup>-</sup>/ CD16<sup>+</sup>/CD56<sup>+</sup> cells. Nonreactive isotype-matched mAb will be used as control.

Aim 1B. Determine whether an SSRI downregulates inflammation in depressed HIV seropositive individuals. *Hypothesis*: SSRI is superior to placebo in decreasing biomarkers of inflammation (IL-6, CRP). Both MDD and HIV infection are associated with elevated levels of pro-inflammatory cytokines (for review see (7, 128-130). Although increased levels of many cytokines, inflammatory and oxidative stress markers were linked to either of those conditions extensive literature review show that IL-6 and CRP are two markers most consistently associated with both MDD and HIV infection. We



Figure 7. Changes in plasma levels of IL-6 in patients treated with aprepitant. IL-6 levels were measured in plasma of 48 patients HIV positive patients enrolled in aprepitant trial. 29 patients received medication (125, 250 or 375 mg per day), 19 received placebo for 14 days. Changes in IL-6 are shown as delta [IL-6] between baseline and after 2 weeks of treatment with aprepitant measured.

propose to use changes in those two markers as a primary outcome of our study. For example in our recent clinical trial with aprepitant, a compound with potential utility as a drug for depression and anti-inflammatory properties in HIV infected subjects, in non-depressed subjects we detected a decrease in plasma levels of IL-6 after 2 weeks of treatment within subjects (p=0.02) and between aprepitant and placebo (p=0.02) (131) (Figure 7). In addition to our primary variables (IL-6 and CRP) associated with inflammation, we will measure several other plasma markers of inflammation in HIV positive depressed subjects receiving SSRI or placebo (see C.4 Further Analyses).

**Secondary Aim.** Determine if improvement in depressive symptoms is associated with improvements in innate immunity and inflammation in HIV seropositive individuals.

Hypothesis: Reduced symptoms of depression after acute (10-week) treatment will correlate with increased

levels of innate immunity (LUNK and intra cellular IFNγ in natural killer cells) and decreased levels of systemic inflammation (IL-6 and CRP).

# C.3.2 Biostatistical Consideration and Analysis Plan

# C.3.2.a Methods and Approach

<u>Primary Aims:</u> For Primary Aims 1A and 1B, participants will provide measures of innate immunity (LUNK and intracellular IFN-γ) and inflammation (IL6 and CRP) at baseline, and at weeks 2, 4, and 10. The measures will be continuously distributed, and we will use linear mixed effects models, probably after log transformation of a response, to estimate the effects of medication group and time on the distribution of the responses across the 10 week period. The explanatory variables in these models will be a binary indicator of medication group, variables representing time effects, together with possible group by time interaction terms. Time will be modeled as a discrete factor. For the covariance structure, we expect that a random intercept model will provide a good fit to the data, and will also compare other possible specifications using BIC comparisons. <u>Secondary Aim:</u> In the Secondary Aim, we will examine relationships between the effects of Escitalopram versus Placebo on depressive symptoms and the effects on the primary biological responses. Hamilton scores will be obtained at baseline and at weeks 2, 4, and 10.

First, we will examine whether participants showing improvement in depression measures are also those showing improvement in primary biological measures. Here, we will calculate change from baseline scores for the Hamilton and for the four immunity measures. For each immunity measure and Hamilton, we will use bivariate mixed effects models to simultaneously model the pattern of depression change scores and immunity change scores across weeks 2 through 10. Here, for each of the four immunity measures, we are modeling the three Hamilton change scores and the three immunity change scores as a six-dimensional response, with explanatory variables of week, medication, and type of response (depression versus immunity). Our hypotheses, that decreases in Hamilton will be associated with increases in innate immunity, and with decreases in inflammation, will be tested by modeling the covariance structure, and testing individual covariances for significant differences from zero. We will perform these analyses separately for the four immunity responses.

Second, we will test whether Escitalopram has direct and indirect effects on the immune responses. The primary analyses (for Aims 1A and 1B) have addressed the total effect of Escitalopram on the four immunity measures. One set of analyses will use the confidence limit approach of MacKinnon et al (135, 136), to test whether changes in Hamilton score at week 2 (and, separately, at week 4) mediate the change in immunity measures at week 10. To obtain a complete picture of the possible mediation effects of depression, we will also perform these analyses using 50% reduction in HAM-D, and HAM-D ≤7, as the measures of the direct effect of Escitalopram on depression. We will perform these analyses on the four innate immunity and inflammation responses separately. These mediation analyses focus on the end of treatment time point. To obtain information on longitudinal mediation across the full period, we will use latent growth curve mediation models (MacKinnon, 2008, 8.10-8.14). These models are similar to the bivariate mixed effects models describe above, but here we include additional regression terms to isolate effects of depression on immunity across time, and random intercepts and slopes for the repeated depression scores and the repeated immunity scores, with the intercept and slope of the immunity response regressed on the intercept and slope of the depression response. MacKinnon (2008) describes how the estimated coefficients of these models can be used to provide estimates and confidence intervals for the indirect and direct effects of Escitalopram on immunity.

# C.3.2.b Power Analysis and Sample Size Calculation for Primary Aims

We use two-sided hypothesis tests, and assume 10% loss to attrition over the 10 weeks. We set an overall alpha level of 5% within the innate immunity and inflammation hypotheses, so each Hypothesis is tested at alpha=0.025. We use the methods of Hedeker et al (122): assuming a within person correlation of 0.6 between visits, we have 80% power to detect a linear group by time effect (from week 0 through week 10) of Cohen's d=0.40 or higher, and 80% power to detect a main effect (from week 2 through week 10) of d=0.4 or higher.

#### C.3.3 Expected Outcomes, Potential Problems and Alternative Approaches

If successful, this trial will advance the field of HIV care by demonstrating the benefit of SSRI treatment on immune system homeostasis, marked by less innate immune suppression and less systemic inflammation, both of which are implicated in HIV pathogenesis. We expect to detect restoration of NK cell functions and decreases in levels of pro inflammatory markers as a result of SSRI treatment. Pro-inflammatory cytokines are thought to play a role in the pathophysiology of depression (4, 7, 86, 132). Although this is not an aim of the present study, data accumulated during our study will allow us to evaluate this relationship along with other patient characteristics (see C.4 Further Analyses). Both depression and HIV are associated with increased plasma levels of IFNy (133, 134) however based on previous observations (42) we expect to see decreased

IFNγ production by stimulated NK cells from HIV+ subjects on cART. We will monitor if SSRI treatment or/and depression improvement will restore IFNγ production. However if we do not detect changes in IFN-γ we will analyze other markers of NK activation and degranulation which are associated with both chronic HIV infection and depression (126) as noted below in C.4. Further Analyses.

We expect to see Immune changes prior to depression improvements suggesting direct SSRI effects on peripheral immune cells. Although unlikely, It is possible that a ceiling effect could be observed and both groups exhibit similar and maximal immune changes at a given time point. If that is the case the frequency of our measures will allow us to study the time course of these immune changes over time and over the time course of depression improvement which will further inform us about SSRI direct effects and depression improvement effects on immunity.

If successful, this rigorously designed clinical trial will advance the field of HIV care by demonstrating the immune benefits of SSRIs among depressed patients with well-controlled viral load – an increasingly prevalent population in the era of modern cART. Many large scale clinical trials encounter challenges with recruitment and retention. We will proactively monitor accrual and retention and should we encounter this challenge, we will initiate a response that will include consultation with the PMHARC Community Advisory Board to discuss recruitment barriers, additional avenues of recruitment and retention strategies. We will also maintain close communications with the Philadelphia Integrated Behavioral Health Initiative which has staff embedded within six of the largest HIV care sites in the city. These staff can help promote recruitment and facilitate retention should we need assistance.

### C.4 Further Analyses

Innate Immunity, Inflammation and Virology: We will also assess the effects of SSRI on other important innate immune cell populations. These responses will be available at baseline and after 2, 4 and 10 weeks of treatment, so they will be analyzed using the approach described above for the primary outcomes of Aim 1. We will evaluate NK receptor expression before and after 10 weeks of SSRI treatment using Flow cytometry assay. Total NK cells will be characterized as CD45<sup>+</sup>/CD3<sup>-</sup>/CD16<sup>+</sup>/CD56<sup>+</sup>. In addition, the expression of the following receptors will be assessed: NKp44, NKp46, NKp30 and CD107 using appropriate antibodies. CD56 bright and dim cells will be also assessed. CD56bright NK cells are associated with cytokine production while CD56 dim are linked to higher cytotoxic activity (137).

In addition to IL-6 and CRP we identified several other markers for further analyses based on the literature and our own immunologic investigations. Specifically, in the aprepitant trial, in addition to IL-6 we also detected a decrease in plasma levels of TNFα and soluble CD163 (sCD163) and decreased expression of Programmed Death 1 (PD-1) receptor on CD4+ cells. PD-1 is known to suppress T cell activation (138). The assays will be done in conjunction with PMHARC Core E. sCD163 and TNF-α will be measured by standard ELISA techniques and PD-1 by flow cytometry. We will use a PD-1 panel established in our laboratory as a part of clinical the trial U01 MH090325 (CD3/CD4/CD8/CD45RO/CD197/CD62L/CD95/PD-1/CD38/HLA-DR). We will also use the monocyte activation/polarization panel which we have developed (CD3/CD14/CD19/CD56/CD16/CD163/CD97/CD312/CD38/HLA-DR). Further we will quantitate expression of CD4, CCR5, and CXCR4 receptors on PBMCs and macrophages to evaluate SSRI effect we observed ex vivo (see C1.9.c). We will measure both fluid phase (plasma) and cellular markers of innate immunity and inflammation using multiplex and flow cytometry technology. These measures will be performed on stored plasma samples and cryopreserved PBMCs.

We expect to find undetectable levels of virus in plasma (<40 copies/ml) in most subjects because all subjects will be on a stable cART regimen. Therefore, data on plasmas viral load will be used primarily for monitoring cART adherence. In contrast, we expect to find low but detectable levels of viral DNA in most subjects. Restoration of NK functions may lead to decreased viral DNA levels. We will analyze if such a decrease is linked to SSRI treatment or improvement of depression in general. We will also establish a repository of plasma and frozen PBMC samples from the 180 depressed HIV+ subjects. This repository will allow us to evaluate other markers associated with depression and/or chronic HIV infection such as oxidative stress (e.g. malondealdedyde), markers of monocyte activation (e.g. neopterin) and any other newly identified molecules during the period of the current study. We will evaluate monocyte activation/polarization profile since we expect that changes in plasma cytokines may affect monocyte polarization which in turn may influence both depression and HIV infection (30-33).

Effects of patient characteristics: Differences in patient demographics (such as age and gender) and characteristics (such as depression severity, levels of life stress, social support, neurocognitive capacity, time since HIV diagnosis, endocrine status, and systemic inflammation level) could potentially moderate the effects of SSRI treatment on our primary outcomes. Some research has suggested that baseline levels of CRP (139), IL-6 and TNF- $\alpha$  (7, 86, 140, 141) and of other biological indicators (7, 86, 132) may influence the effects of

SSRI on depression. We will perform a series of moderator analyses (142) to address these questions. The potential moderators will be included as main effects and as interactions with group in the analyses described above for the primary responses. We will use multivariate analyses analogous to the univariate analyses to examine SSRI effects on a wider range of biological responses to include endocrine hormones (cortisol, ACTH, DHEA), as well as the flow cytometry panels noted above.

**C.5 Missing Data and Nonadherence** For the primary analyses described above, premature discontinuation from treatment and occasional missing weekly appointments will lead to incomplete data. The mixed effects models for Aim 1, Hypothesis 1 described above can make use of all available data provided by subjects, but the inferences drawn from them will be unaffected by the missing data only if the missing data can be regarded as ignorable. For the other primary responses, dropouts will not provide any responses, so the basic models require ignorable dropout. To assess the sensitivity of our analyses to this assumption, we will also use selection models (143) to examine the effects of missing data: we will explicitly model the probability of premature discontinuation at a time point as a function of baseline characteristics and responses at previous time points, using a logistic regression model. For the longitudinal analyses of Aim 1, Hypothesis 1, these probabilities will provide time varying (inverse) weights for reruns of the primary analysis. For the other primary hypotheses, the overall probability of dropout will be used as a weight, and incorporated into a weighted analysis of these hypotheses. We will perform these analyses in a range of assumptions on the dropout process and assess the sensitivity of results to them. To account for possible non-adherence to assigned intervention, we will use self-report of pill ingestion and MEMS caps, as well as RNA viral load for cART. We will use the methods of Nagelkerke et al (144, 145), to obtain estimates of the intervention effect in a population compliant with treatment i.e. the Complier Average Causal Effect (CACE).

**C.6 Data Management** Data will be gathered using an internet-based direct-entry data system developed and used over the last ten years by the U Penn Center for Studies on Addictions in the Department of Psychiatry. Interview data and self-report data are entered directly onto computers at the research sites by research technicians and study subjects respectively. Field validation (e.g., no out-of-range or otherwise invalid responses will be accepted) and form validation (e.g., logically impossible responses to different questions will not be accepted) are built into this entry process. Data are transmitted (128-bit encrypted form) over the Internet to the DMU servers. After online reviews, the data are archived on secure servers located in the U Penn School of Medicine Data Center. No identifying information is stored on the DMU servers. Certain DMU staff members have permission to modify the archived data. Audit logs record any modification to the original entry. Password protection allows members of the research team appropriate levels of data access.

### **References Cited**

- 1. Ciesla JA, Roberts JE. Meta-analysis of the relationship between HIV infection and risk for depressive disorders. The American journal of psychiatry. 2001;158(5):725-30. PubMed PMID: 11329393.
- 2. Ownby R, Jacobs, RJ, Waldrop-Valverde, D, Gould, F. Depression Care and Prevalence in HIV-positive individuals. Neurobehavioral HIV Medicine. 2010(2):73-83.
- 3. Zorrilla EP, Luborsky L, McKay JR, Rosenthal R, Houldin A, Tax A, McCorkle R, Seligman DA, Schmidt K. The relationship of depression and stressors to immunological assays: a meta-analytic review. Brain, behavior, and immunity. 2001;15(3):199-226. doi: 10.1006/brbi.2000.0597. PubMed PMID: 11566046.
- 4. Irwin MR, Miller AH. Depressive disorders and immunity: 20 years of progress and discovery. Brain, behavior, and immunity. 2007;21(4):374-83. doi: 10.1016/j.bbi.2007.01.010. PubMed PMID: 17360153.
- 5. Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosomatic medicine. 2009;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. PubMed PMID: 19188531.
- 6. Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biological psychiatry. 2010;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. PubMed PMID: 20015486.
- 7. Blume J, Douglas SD, Evans DL. Immune suppression and immune activation in depression. Brain, behavior, and immunity. 2011;25(2):221-9. doi: 10.1016/j.bbi.2010.10.008. PubMed PMID: 20955778; PubMed Central PMCID: PMC3025086.
- 8. Hannestad J, DellaGioia N, Bloch M. The effect of antidepressant medication treatment on serum levels of inflammatory cytokines: a meta-analysis. Neuropsychopharmacology. 2011;36(12):2452-9. doi: 10.1038/npp.2011.132. PubMed PMID: 21796103; PubMed Central PMCID: PMC3194072.
- 9. Hiles SA, Baker AL, de Malmanche T, Attia J. Interleukin-6, C-reactive protein and interleukin-10 after antidepressant treatment in people with depression: a meta-analysis. Psychological medicine. 2012;42(10):2015-26. doi: 10.1017/S0033291712000128. PubMed PMID: 22336436.
- 10. Evans DL, Charney DS, Lewis L, Golden RN, Gorman JM, Krishnan KR, Nemeroff CB, Bremner JD, Carney RM, Coyne JC, Delong MR, Frasure-Smith N, Glassman AH, Gold PW, Grant I, Gwyther L, Ironson G, Johnson RL, Kanner AM, Katon WJ, Kaufmann PG, Keefe FJ, Ketter T, Laughren TP, Leserman J, Lyketsos CG, McDonald WM, McEwen BS, Miller AH, Musselman D, O'Connor C, Petitto JM, Pollock BG, Robinson RG, Roose SP, Rowland J, Sheline Y, Sheps DS, Simon G, Spiegel D, Stunkard A, Sunderland T, Tibbits P, Jr., Valvo WJ. Mood disorders in the medically ill: scientific review and recommendations. Biological psychiatry. 2005;58(3):175-89. doi: 10.1016/j.biopsych.2005.05.001. PubMed PMID: 16084838.
- 11. Schleifer SJ, Keller SE, Bond RN, Cohen J, Stein M. Major depressive disorder and immunity. Role of age, sex, severity, and hospitalization. Archives of general psychiatry. 1989;46(1):81-7. PubMed PMID: 2562915.
- 12. Evans DL, Leserman J, Pedersen CA, Golden RN, Lewis MH, Folds JA, Ozer H. Immune correlates of stress and depression. Psychopharmacology bulletin. 1989;25(3):319-24. PubMed PMID: 2697005.
- 13. Sephton SE, Kraemer HC, Neri E, Stites DP, Weissbecker I, Spiegel D. Improving methods of assessing natural killer cell cytotoxicity. International journal of methods in psychiatric research. 2006;15(1):12-21. PubMed PMID: 16676682.
- 14. Phillips MI, Evans D. Neuroimmunology. San Diego: Academic Press; 1995. xx, 434 p. p.
- 15. Rabin B. Stress, Immune Function and Health: The Connection. Rabin B, editor. New York: Wiley-Liss and Sons; 1999.
- 16. Glaser R, Rabin B, Chesney M, Cohen S, Natelson B. Stress-induced immunomodulation: implications for infectious diseases? JAMA. 1999;281(24):2268-70. PubMed PMID: 10386538.
- 17. Kiecolt-Glaser JK, Glaser R. Depression and immune function: central pathways to morbidity and mortality. Journal of psychosomatic research. 2002;53(4):873-6. PubMed PMID: 12377296.
- 18. Raison CL, Miller AH. The neuroimmunology of stress and depression. Seminars in clinical neuropsychiatry. 2001;6(4):277-94. PubMed PMID: 11607923.
- 19. Ironson G, Hayward H. Do positive psychosocial factors predict disease progression in HIV-1? A review of the evidence. Psychosomatic medicine. 2008;70(5):546-54. doi: 10.1097/PSY.0b013e318177216c. PubMed PMID: 18541905; PubMed Central PMCID: PMC2614870.
- 20. Burack JH, Barrett DC, Stall RD, Chesney MA, Ekstrand ML, Coates TJ. Depressive symptoms and CD4 lymphocyte decline among HIV-infected men. JAMA. 1993;270(21):2568-73. PubMed PMID: 7901433.
- 21. Evans DL, Ten Have TR, Douglas SD, Gettes DR, Morrison M, Chiappini MS, Brinker-Spence P, Job C, Mercer DE, Wang YL, Cruess D, Dube B, Dalen EA, Brown T, Bauer R, Petitto JM. Association of depression with viral load, CD8 T lymphocytes, and natural killer cells in women with HIV infection. The American journal of psychiatry. 2002;159(10):1752-9. PubMed PMID: 12359683.

- 22. Ickovics JR, Hamburger ME, Vlahov D, Schoenbaum EE, Schuman P, Boland RJ, Moore J, Group HIVERS. Mortality, CD4 cell count decline, and depressive symptoms among HIV-seropositive women: longitudinal analysis from the HIV Epidemiology Research Study. JAMA 2001;285(11):1466-74. PubMed PMID: 11255423.
- 23. Lyketsos CG, Hoover DR, Guccione M, Dew MA, Wesch JE, Bing EG, Treisman GJ. Changes in depressive symptoms as AIDS develops. The Multicenter AIDS Cohort Study. The American journal of psychiatry. 1996;153(11):1430-7. PubMed PMID: 8890676.
- Mayne TJ, Vittinghoff E, Chesney MA, Barrett DC, Coates TJ. Depressive affect and survival among gay and bisexual men infected with HIV. Archives of internal medicine. 1996;156(19):2233-8. PubMed PMID: 8885823.
- 25. Page-Shafer K, Delorenze GN, Satariano WA, Winkelstein W, Jr. Comorbidity and survival in HIV-infected men in the San Francisco Men's Health Survey. Annals of epidemiology. 1996;6(5):420-30. PubMed PMID: 8915473.
- 26. Leserman J. Role of depression, stress, and trauma in HIV disease progression. Psychosomatic medicine. 2008;70(5):539-45. doi: 10.1097/PSY.0b013e3181777a5f. PubMed PMID: 18519880.
- 27. Temoshok LR, Wald RL, Synowski S, Garzino-Demo A. Coping as a multisystem construct associated with pathways mediating HIV-relevant immune function and disease progression. Psychosomatic medicine. 2008;70(5):555-61. doi: 10.1097/PSY.0b013e318177354f. PubMed PMID: 18519884.
- 28. Patterson TL, Shaw WS, Semple SJ, Cherner M, McCutchan JA, Atkinson JH, Grant I, Nannis E, Group HIVNRC. Relationship of psychosocial factors to HIV disease progression. Annals of behavioral medicine: a publication of the Society of Behavioral Medicine. 1996;18(1):30-9. doi: 10.1007/BF02903937. PubMed PMID: 24203641.
- 29. Stein M, Miller AH, Trestman RL. Depression, the immune system, and health and illness. Findings in search of meaning. Archives of general psychiatry. 1991;48(2):171-7. PubMed PMID: 1671201.
- 30. Herbert TB, Cohen S. Depression and immunity: a meta-analytic review. Psychological bulletin. 1993;113(3):472-86. PubMed PMID: 8316610.
- 31. Evans DL, Folds JD, Petitto JM, Golden RN, Pedersen CA, Corrigan M, Gilmore JH, Silva SG, Quade D, Ozer H. Circulating natural killer cell phenotypes in men and women with major depression. Relation to cytotoxic activity and severity of depression. Archives of general psychiatry. 1992;49(5):388-95. PubMed PMID: 1534002.
- 32. Fauci AS, Mavilio D, Kottilil S. NK cells in HIV infection: paradigm for protection or targets for ambush. Nature reviews Immunology. 2005;5(11):835-43. doi: 10.1038/nri1711. PubMed PMID: 16239902.
- 33. Oliva A, Kinter AL, Vaccarezza M, Rubbert A, Catanzaro A, Moir S, Monaco J, Ehler L, Mizell S, Jackson R, Li Y, Romano JW, Fauci AS. Natural killer cells from human immunodeficiency virus (HIV)-infected individuals are an important source of CC-chemokines and suppress HIV-1 entry and replication in vitro. The Journal of clinical investigation. 1998;102(1):223-31. doi: 10.1172/JCI2323. PubMed PMID: 9649576; PubMed Central PMCID: PMC509084.
- 34. Poli G, Fauci AS. The effect of cytokines and pharmacologic agents on chronic HIV infection. AIDS research and human retroviruses. 1992;8(2):191-7. PubMed PMID: 1540407.
- 35. Cocchi F, DeVico AL, Garzino-Demo A, Arya SK, Gallo RC, Lusso P. Identification of RANTES, MIP-1 alpha, and MIP-1 beta as the major HIV-suppressive factors produced by CD8+ T cells. Science. 1995;270(5243):1811-5. PubMed PMID: 8525373.
- 36. Chehimi J, Starr SE, Frank I, Rengaraju M, Jackson SJ, Llanes C, Kobayashi M, Perussia B, Young D, Nickbarg E, et al. Natural killer (NK) cell stimulatory factor increases the cytotoxic activity of NK cells from both healthy donors and human immunodeficiency virus-infected patients. The Journal of experimental medicine. 1992;175(3):789-96. PubMed PMID: 1346797; PubMed Central PMCID: PMC2119140.
- 37. Bandyopadhyay S, Ziegner U, Campbell DE, Miller DS, Hoxie JA, Starr SE. Natural killer cell-mediated lysis of T cell lines chronically infected with HIV-1. Clinical and experimental immunology. 1990;79(3):430-5. PubMed PMID: 1969336; PubMed Central PMCID: PMC1534966.
- 38. Fauci AS, Pantaleo G, Stanley S, Weissman D. Immunopathogenic mechanisms of HIV infection. Annals of internal medicine. 1996;124(7):654-63. PubMed PMID: 8607594.
- 39. Ferbas J. Perspectives on the role of CD8+ cell suppressor factors and cytotoxic T lymphocytes during HIV infection. AIDS research and human retroviruses. 1998;14 Suppl 2:S153-60. PubMed PMID: 9672233.
- 40. Barker E, Bossart KN, Levy JA. Primary CD8+ cells from HIV-infected individuals can suppress productive infection of macrophages independent of beta-chemokines. Proceedings of the National Academy of Sciences of the United States of America. 1998;95(4):1725-9. PubMed PMID: 9465084; PubMed Central PMCID: PMC19166.
- 41. Douglas SD, Durako SJ, Tustin NB, Houser J, Muenz L, Starr SE, Wilson C, Adolescent Medicine HIVARN. Natural killer cell enumeration and function in HIV-infected and high-risk uninfected adolescents.

- AIDS research and human retroviruses. 2001;17(6):543-52. doi: 10.1089/08892220151126643. PubMed PMID: 11350668.
- 42. Azzoni L, Papasavvas E, Chehimi J, Kostman JR, Mounzer K, Ondercin J, Perussia B, Montaner LJ. Sustained impairment of IFN-gamma secretion in suppressed HIV-infected patients despite mature NK cell recovery: evidence for a defective reconstitution of innate immunity. Journal of immunology. 2002;168(11):5764-70. PubMed PMID: 12023377.
- 43. Fortis C, Tasca S, Capiluppi B, Tambussi G. Natural killer cell function in HIV-1 infected patients. Journal of biological regulators and homeostatic agents. 2002;16(1):30-2. PubMed PMID: 12003170.
- 44. Chehimi J, Azzoni L, Farabaugh M, Creer SA, Tomescu C, Hancock A, Mackiewicz A, D'Alessandro L, Ghanekar S, Foulkes AS, Mounzer K, Kostman J, Montaner LJ. Baseline viral load and immune activation determine the extent of reconstitution of innate immune effectors in HIV-1-infected subjects undergoing antiretroviral treatment. Journal of immunology. 2007;179(4):2642-50. PubMed PMID: 17675528.
- 45. Goodier MR, Imami N, Moyle G, Gazzard B, Gotch F. Loss of the CD56hiCD16- NK cell subset and NK cell interferon-gamma production during antiretroviral therapy for HIV-1: partial recovery by human growth hormone. Clinical and experimental immunology. 2003;134(3):470-6. PubMed PMID: 14632753; PubMed Central PMCID: PMC1808890.
- 46. Lichtfuss GF, Cheng WJ, Farsakoglu Y, Paukovics G, Rajasuriar R, Velayudham P, Kramski M, Hearps AC, Cameron PU, Lewin SR, Crowe SM, Jaworowski A. Virologically suppressed HIV patients show activation of NK cells and persistent innate immune activation. Journal of immunology. 2012;189(3):1491-9. doi: 10.4049/jimmunol.1200458. PubMed PMID: 22745371.
- 47. French MA, King MS, Tschampa JM, da Silva BA, Landay AL. Serum immune activation markers are persistently increased in patients with HIV infection after 6 years of antiretroviral therapy despite suppression of viral replication and reconstitution of CD4+ T cells. Journal of infectious diseases. 2009;200(8):1212-5. PubMed PMID: 19728788.
- 48. Sandler NG, Wand H, Roque A, Law M, Nason MC, Nixon DE, Pedersen C, Ruxrungtham K, Lewin SR, Emery S, Neaton JD, Brenchley JM, Deeks SG, Sereti I, Douek DC, Group ISS. Plasma levels of soluble CD14 independently predict mortality in HIV infection. The Journal of infectious diseases. 2011;203(6):780-90. doi: 10.1093/infdis/jig118. PubMed PMID: 21252259; PubMed Central PMCID: PMC3071127.
- 49. Rajasuriar R, Khoury G, Kamarulzaman A, French MA, Cameron PU, Lewin SR. Persistent immune activation in chronic HIV infection: do any interventions work? AIDS. 2013;27(8):1199-208. doi: 10.1097/QAD.0b013e32835ecb8b. PubMed PMID: 23324661.
- 50. Stein JH, Hsue PY. Inflammation, immune activation, and CVD risk in individuals with HIV infection. JAMA: the journal of the American Medical Association. 2012;308(4):405-6. PubMed PMID: 22820794.
- 51. Subramanian S, Tawakol A, Burdo TH, Abbara S, Wei J, Vijayakumar J, Corsini E, Abdelbaky A, Zanni MV, Hoffmann U, Williams KC, Lo J, Grinspoon SK. Arterial inflammation in patients with HIV. JAMA: the journal of the American Medical Association. 2012;308(4):379-86. PubMed PMID: 22820791.
- 52. Kulpa DA, Brehm JH, Fromentin R, Cooper A, Cooper C, Ahlers J, Chomont N, Sekaly RP. The immunological synapse: the gateway to the HIV reservoir. Immunological reviews. 2013;254(1):305-25. doi: 10.1111/imr.12080. PubMed PMID: 23772628; PubMed Central PMCID: PMC3707302.
- 53. Porichis F, Hart MG, Zupkosky J, Barblu L, Kwon DS, McMullen A, Brennan T, Ahmed R, Freeman GJ, Kavanagh DG, Kaufmann DE. Differential impact of PD-1 and/or interleukin-10 blockade on HIV-1-specific CD4 T cell and antigen-presenting cell functions. J Virol. 2014;88(5):2508-18. doi: 10.1128/JVI.02034-13. PubMed PMID: 24352453; PubMed Central PMCID: PMC3958087.
- 54. Barouch DH, Deeks SG. Immunologic strategies for HIV-1 remission and eradication. Science. 2014;345(6193):169-74. doi: 10.1126/science.1255512. PubMed PMID: 25013067; PubMed Central PMCID: PMC4096716.
- 55. Zeng M, Haase AT, Schacker TW. Lymphoid tissue structure and HIV-1 infection: life or death for T cells. Trends in immunology. 2012;33(6):306-14. doi: 10.1016/j.it.2012.04.002. PubMed PMID: 22613276.
- 56. Delgado PL, Price LH, Miller HL, Salomon RM, Aghajanian GK, Heninger GR, Charney DS. Serotonin and the neurobiology of depression. Effects of tryptophan depletion in drug-free depressed patients. Archives of general psychiatry. 1994;51(11):865-74. PubMed PMID: 7944875.
- 57. Mann JJ. The medical management of depression. The New England journal of medicine. 2005;353(17):1819-34. doi: 10.1056/NEJMra050730. PubMed PMID: 16251538.
- 58. Mossner R, Lesch KP. Role of serotonin in the immune system and in neuroimmune interactions. Brain, behavior, and immunity. 1998;12(4):249-71. doi: 10.1006/brbi.1998.0532. PubMed PMID: 10080856.
- 59. Young MR, Matthews JP. Serotonin regulation of T-cell subpopulations and of macrophage accessory function. Immunology. 1995;84(1):148-52. PubMed PMID: 7890297; PubMed Central PMCID: PMC1415171.

- 60. Hellstrand K, Hermodsson S. Enhancement of human natural killer cell cytotoxicity by serotonin: role of non-T/CD16+ NK cells, accessory monocytes, and 5-HT1A receptors. Cellular immunology. 1990;127(1):199-214. PubMed PMID: 2138518.
- 61. Mizruchin A, Gold I, Krasnov I, Livshitz G, Shahin R, Kook AI. Comparison of the effects of dopaminergic and serotonergic activity in the CNS on the activity of the immune system. Journal of neuroimmunology. 1999;101(2):201-4. PubMed PMID: 10580803.
- 62. Dustin ML, Colman DR. Neural and immunological synaptic relations. Science. 2002;298(5594):785-9. doi: 10.1126/science.1076386. PubMed PMID: 12399580.
- 63. Jackson JC, Walker RF, Brooks WH, Roszman TL. Specific uptake of serotonin by murine macrophages. Life sciences. 1988;42(17):1641-50. PubMed PMID: 2452944.
- 64. Finocchiaro LM, Arzt ES, Fernandez-Castelo S, Criscuolo M, Finkielman S, Nahmod VE. Serotonin and melatonin synthesis in peripheral blood mononuclear cells: stimulation by interferon-gamma as part of an immunomodulatory pathway. Journal of interferon research. 1988;8(6):705-16. PubMed PMID: 3148005.
- 65. Faraj BA, Olkowski ZL, Jackson RT. Expression of a high-affinity serotonin transporter in human lymphocytes. International journal of immunopharmacology. 1994;16(7):561-7. PubMed PMID: 7928004.
- Aune TM, Kelley KA, Ranges GE, Bombara MP. Serotonin-activated signal transduction via serotonin receptors on Jurkat cells. Journal of immunology. 1990;145(6):1826-31. PubMed PMID: 2144010.
- 67. Choquet D, Korn H. Dual effects of serotonin on a voltage-gated conductance in lymphocytes. Proceedings of the National Academy of Sciences of the United States of America. 1988;85(12):4557-61. PubMed PMID: 3260036; PubMed Central PMCID: PMC280470.
- 68. Fargin A, Raymond JR, Lohse MJ, Kobilka BK, Caron MG, Lefkowitz RJ. The genomic clone G-21 which resembles a beta-adrenergic receptor sequence encodes the 5-HT1A receptor. Nature. 1988;335(6188):358-60. doi: 10.1038/335358a0. PubMed PMID: 3138543.
- 69. Hellstrand K, Hermodsson S. Role of serotonin in the regulation of human natural killer cell cytotoxicity. Journal of immunology. 1987;139(3):869-75. PubMed PMID: 2439597.
- 70. Aune TM, Golden HW, McGrath KM. Inhibitors of serotonin synthesis and antagonists of serotonin 1A receptors inhibit T lymphocyte function in vitro and cell-mediated immunity in vivo. Journal of immunology. 1994;153(2):489-98. PubMed PMID: 8021490.
- 71. Evans DL, Lynch KG, Benton T, Dube B, Gettes DR, Tustin NB, Lai JP, Metzger D, Douglas SD. Selective serotonin reuptake inhibitor and substance P antagonist enhancement of natural killer cell innate immunity in human immunodeficiency virus/acquired immunodeficiency syndrome. Biological psychiatry. 2008;63(9):899-905. Epub 2007/10/20. doi: S0006-3223(07)00820-7 [pii]
- 10.1016/j.biopsych.2007.08.012. PubMed PMID: 17945197; PubMed Central PMCID: PMC2845393.
- 72. Benton T, Lynch K, Dube B, Gettes DR, Tustin NB, Ping Lai J, Metzger DS, Blume J, Douglas SD, Evans DL. Selective serotonin reuptake inhibitor suppression of HIV infectivity and replication. Psychosomatic medicine. 2010;72(9):925-32. Epub 2010/10/16. doi: PSY.0b013e3181f883ce [pii]
- 10.1097/PSY.0b013e3181f883ce. PubMed PMID: 20947783; PubMed Central PMCID: PMC2978281.
- 73. Frank MG, Hendricks SE, Johnson DR, Wieseler JL, Burke WJ. Antidepressants augment natural killer cell activity: in vivo and in vitro. Neuropsychobiology. 1999;39(1):18-24. doi: 26555. PubMed PMID: 9892855.
- 74. Kook AI, Mizruchin A, Odnopozov N, Gershon H, Segev Y. Depression and immunity: the biochemical interrelationship between the central nervous system and the immune system. Biological psychiatry. 1995;37(11):817-9. doi: 10.1016/0006-3223(95)00038-I. PubMed PMID: 7647167.
- 75. Irwin M, Lacher U, Caldwell C. Depression and reduced natural killer cytotoxicity: a longitudinal study of depressed patients and control subjects. Psychological medicine. 1992;22(4):1045-50. PubMed PMID: 1488477.
- 76. Cruess DG, Douglas SD, Petitto JM, Have TT, Gettes D, Dube B, Cary M, Evans DL. Association of resolution of major depression with increased natural killer cell activity among HIV-seropositive women. The American journal of psychiatry. 2005;162(11):2125-30. doi: 10.1176/appi.ajp.162.11.2125. PubMed PMID: 16263853.
- 77. Hofmann B, Nishanian P, Nguyen T, Liu M, Fahey JL. Restoration of T-cell function in HIV infection by reduction of intracellular cAMP levels with adenosine analogues. AIDS. 1993;7(5):659-64. PubMed PMID: 8391271.
- 78. Hofmann B, Afzelius P, Iversen J, Kronborg G, Aabech P, Benfield T, Dybkjaer E, Nielsen JO. Buspirone, a serotonin receptor agonist, increases CD4 T-cell counts and modulates the immune system in HIV-seropositive subjects. AIDS. 1996;10(12):1339-47. PubMed PMID: 8902062.
- 79. Eugen-Olsen J, Afzelius P, Andresen L, Iversen J, Kronborg G, Aabech P, Nielsen JO, Hofmann B. Serotonin modulates immune function in T cells from HIV-seropositive subjects. Clinical immunology and immunopathology. 1997;84(2):115-21. PubMed PMID: 9245541.

- 80. Gordon J, Barnes NM. Lymphocytes transport serotonin and dopamine: agony or ecstasy? Trends in immunology. 2003;24(8):438-43. PubMed PMID: 12909457.
- 81. O'Connell PJ, Wang X, Leon-Ponte M, Griffiths C, Pingle SC, Ahern GP. A novel form of immune signaling revealed by transmission of the inflammatory mediator serotonin between dendritic cells and T cells. Blood. 2006;107(3):1010-7. doi: 10.1182/blood-2005-07-2903. PubMed PMID: 16223770; PubMed Central PMCID: PMC1895901.
- 82. Letendre SL, Marquie-Beck J, Ellis RJ, Woods SP, Best B, Clifford DB, Collier AC, Gelman BB, Marra C, McArthur JC, McCutchan JA, Morgello S, Simpson D, Alexander TJ, Durelle J, Heaton R, Grant I, Group C. The role of cohort studies in drug development: clinical evidence of antiviral activity of serotonin reuptake inhibitors and HMG-CoA reductase inhibitors in the central nervous system. Journal of neuroimmune pharmacology: the official journal of the Society on NeuroImmune Pharmacology. 2007;2(1):120-7. doi: 10.1007/s11481-006-9054-y. PubMed PMID: 18040835.
- 83. Liu D, Wang Z, Liu S, Wang F, Zhao S, Hao A. Anti-inflammatory effects of fluoxetine in lipopolysaccharide(LPS)-stimulated microglial cells. Neuropharmacology. 2011;61(4):592-9. doi: 10.1016/i.neuropharm.2011.04.033. PubMed PMID: 21575647.
- 84. Tynan RJ, Weidenhofer J, Hinwood M, Cairns MJ, Day TA, Walker FR. A comparative examination of the anti-inflammatory effects of SSRI and SNRI antidepressants on LPS stimulated microglia. Brain, behavior, and immunity. 2012;26(3):469-79. doi: 10.1016/j.bbi.2011.12.011. PubMed PMID: 22251606.
- 85. Maneglier B, Guillemin GJ, Clayette P, Rogez-Kreuz C, Brew BJ, Dormont D, Advenier C, Therond P, Spreux-Varoquaux O. Serotonin decreases HIV-1 replication in primary cultures of human macrophages through 5-HT(1A) receptors. British journal of pharmacology. 2008;154(1):174-82. doi: 10.1038/bjp.2008.80. PubMed PMID: 18332855; PubMed Central PMCID: PMC2438982.
- 86. Miller AH, Maletic V, Raison CL. Inflammation and its discontents: the role of cytokines in the pathophysiology of major depression. Biological psychiatry. 2009;65(9):732-41. doi:
- 10.1016/j.biopsych.2008.11.029. PubMed PMID: 19150053; PubMed Central PMCID: PMC2680424.
- 87. Vogelzangs N, Duivis HE, Beekman AT, Kluft C, Neuteboom J, Hoogendijk W, Smit JH, de Jonge P, Penninx BW. Association of depressive disorders, depression characteristics and antidepressant medication with inflammation. Translational psychiatry. 2012;2:e79. doi: 10.1038/tp.2012.8. PubMed PMID: 22832816; PubMed Central PMCID: PMC3309556.
- 88. O'Brien SM, Scott LV, Dinan TG. Antidepressant therapy and C-reactive protein levels. The British journal of psychiatry: the journal of mental science. 2006;188:449-52. doi: 10.1192/bjp.bp.105.011015. PubMed PMID: 16648531.
- 89. Sluzewska A, Rybakowski JK, Laciak M, Mackiewicz A, Sobieska M, Wiktorowicz K. Interleukin-6 serum levels in depressed patients before and after treatment with fluoxetine. Annals of the New York Academy of Sciences. 1995;762:474-6. PubMed PMID: 7668562.
- 90. Basterzi AD, Aydemir C, Kisa C, Aksaray S, Tuzer V, Yazici K, Goka E. IL-6 levels decrease with SSRI treatment in patients with major depression. Human psychopharmacology. 2005;20(7):473-6. doi: 10.1002/hup.717. PubMed PMID: 16158446.
- 91. Leo R, Di Lorenzo G, Tesauro M, Razzini C, Forleo GB, Chiricolo G, Cola C, Zanasi M, Troisi A, Siracusano A, Lauro R, Romeo F. Association between enhanced soluble CD40 ligand and proinflammatory and prothrombotic states in major depressive disorder: pilot observations on the effects of selective serotonin reuptake inhibitor therapy. The Journal of clinical psychiatry. 2006;67(11):1760-6. PubMed PMID: 17196057.
- 92. Tuglu C, Kara SH, Caliyurt O, Vardar E, Abay E. Increased serum tumor necrosis factor-alpha levels and treatment response in major depressive disorder. Psychopharmacology. 2003;170(4):429-33. doi: 10.1007/s00213-003-1566-z. PubMed PMID: 12955291.
- 93. Sutcigil L, Oktenli C, Musabak U, Bozkurt A, Cansever A, Uzun O, Sanisoglu SY, Yesilova Z, Ozmenler N, Ozsahin A, Sengul A. Pro- and anti-inflammatory cytokine balance in major depression: effect of sertraline therapy. Clinical & developmental immunology. 2007;2007:76396. doi: 10.1155/2007/76396. PubMed PMID: 18317531; PubMed Central PMCID: PMC2248234.
- 94. Pizzi C, Mancini S, Angeloni L, Fontana F, Manzoli L, Costa GM. Effects of selective serotonin reuptake inhibitor therapy on endothelial function and inflammatory markers in patients with coronary heart disease. Clinical pharmacology and therapeutics. 2009;86(5):527-32. doi: 10.1038/clpt.2009.121. PubMed PMID: 19641491.
- 95. Elliott AJ, Uldall KK, Bergam K, Russo J, Claypoole K, Roy-Byrne PP. Randomized, placebo-controlled trial of paroxetine versus imipramine in depressed HIV-positive outpatients. The American journal of psychiatry. 1998;155(3):367-72. PubMed PMID: 9501747.
- 96. Rabkin JG, Wagner GJ, Rabkin R. Fluoxetine treatment for depression in patients with HIV and AIDS: a randomized, placebo-controlled trial. The American journal of psychiatry. 1999;156(1):101-7. PubMed PMID: 9892304.

- 97. Zisook S, Peterkin J, Goggin KJ, Sledge P, Atkinson JH, Grant I. Treatment of major depression in HIV-seropositive men. HIV Neurobehavioral Research Center Group. The Journal of clinical psychiatry. 1998;59(5):217-24. PubMed PMID: 9632030.
- 98. Hoare J, Carey P, Joska JA, Carrara H, Sorsdahl K, Stein DJ. Escitalopram treatment of depression in human immunodeficiency virus/acquired immunodeficiency syndrome: a randomized, double-blind, placebo-controlled study. The Journal of nervous and mental disease. 2014;202(2):133-7. doi: 10.1097/NMD.000000000000082. PubMed PMID: 24469525.
- 99. Rabkin JG, Wagner GJ, McElhiney MC, Rabkin R, Lin SH. Testosterone versus fluoxetine for depression and fatigue in HIV/AIDS: a placebo-controlled trial. Journal of clinical psychopharmacology. 2004;24(4):379-85. PubMed PMID: 15232328.
- 100. Perkins DO, Stern RA, Golden RN, Murphy C, Naftolowitz D, Evans DL. Mood disorders in HIV infection: prevalence and risk factors in a nonepicenter of the AIDS epidemic. The American journal of psychiatry. 1994;151(2):233-6. PubMed PMID: 8296895.
- 101. Morrison MF, Petitto JM, Ten Have T, Gettes DR, Chiappini MS, Weber AL, Brinker-Spence P, Bauer RM, Douglas SD, Evans DL. Depressive and anxiety disorders in women with HIV infection. The American journal of psychiatry. 2002;159(5):789-96. PubMed PMID: 11986133.
- 102. Evans DL, Leserman J, Perkins DO, Stern RA, Murphy C, Tamul K, Liao D, van der Horst CM, Hall CD, Folds JD, et al. Stress-associated reductions of cytotoxic T lymphocytes and natural killer cells in asymptomatic HIV infection. The American journal of psychiatry. 1995;152(4):543-50. PubMed PMID: 7694902.
- 103. Leserman J, Petitto JM, Perkins DO, Folds JD, Golden RN, Evans DL. Severe stress, depressive symptoms, and changes in lymphocyte subsets in human immunodeficiency virus-infected men. A 2-year follow-up study. Archives of general psychiatry. 1997;54(3):279-85. PubMed PMID: 9075469.
- 104. Evans DL, Leserman J, Perkins DO, Stern RA, Murphy C, Zheng B, Gettes D, Longmate JA, Silva SG, van der Horst CM, Hall CD, Folds JD, Golden RN, Petitto JM. Severe life stress as a predictor of early disease progression in HIV infection. The American journal of psychiatry. 1997;154(5):630-4. PubMed PMID: 9137117.
- 105. Leserman J, Jackson ED, Petitto JM, Golden RN, Silva SG, Perkins DO, Cai J, Folds JD, Evans DL. Progression to AIDS: the effects of stress, depressive symptoms, and social support. Psychosomatic medicine. 1999;61(3):397-406. PubMed PMID: 10367622.
- 106. Leserman J, Petitto JM, Gu H, Gaynes BN, Barroso J, Golden RN, Perkins DO, Folds JD, Evans DL. Progression to AIDS, a clinical AIDS condition and mortality: psychosocial and physiological predictors. Psychological medicine. 2002;32(6):1059-73. PubMed PMID: 12214787.
- 107. Ickovics JR, Milan S, Boland R, Schoenbaum E, Schuman P, Vlahov D, Group HIVERS. Psychological resources protect health: 5-year survival and immune function among HIV-infected women from four US cities. AIDS. 2006;20(14):1851-60. doi: 10.1097/01.aids.0000244204.95758.15. PubMed PMID: 16954726.
- 108. Antinori A, Arendt G, Becker JT, Brew BJ, Byrd DA, Cherner M, Clifford DB, Cinque P, Epstein LG, Goodkin K, Gisslen M, Grant I, Heaton RK, Joseph J, Marder K, Marra CM, McArthur JC, Nunn M, Price RW, Pulliam L, Robertson KR, Sacktor N, Valcour V, Wojna VE. Updated research nosology for HIV-associated neurocognitive disorders. Neurology. 2007;69(18):1789-99. doi: 10.1212/01.WNL.0000287431.88658.8b. PubMed PMID: 17914061.
- 109. Cipriani A, Furukawa TA, Salanti G, Geddes JR, Higgins JP, Churchill R, Watanabe N, Nakagawa A, Omori IM, McGuire H, Tansella M, Barbui C. Comparative efficacy and acceptability of 12 new-generation antidepressants: a multiple-treatments meta-analysis. Lancet. 2009;373(9665):746-58. doi: 10.1016/S0140-6736(09)60046-5. PubMed PMID: 19185342.
- 110. Dohrenwend BS, Krasnoff L, Askenasy AR, Dohrenwend BP. Exemplification of a method for scaling life events: the Peri Life Events Scale. Journal of health and social behavior. 1978;19(2):205-29. PubMed PMID: 681735.
- 111. Grant I, Franklin DR, Jr., Deutsch R, Woods SP, Vaida F, Ellis RJ, Letendre SL, Marcotte TD, Atkinson JH, Collier AC, Marra CM, Clifford DB, Gelman BB, McArthur JC, Morgello S, Simpson DM, McCutchan JA, Abramson I, Gamst A, Fennema-Notestine C, Smith DM, Heaton RK, Group C. Asymptomatic HIV-associated neurocognitive impairment increases risk for symptomatic decline. Neurology. 2014;82(23):2055-62. doi: 10.1212/WNL.0000000000000492. PubMed PMID: 24814848.
- 112. Cheulune G, Heaton RK, Lehman RA. Advances in Clinical Neuropsychology. New York: Plenum Press; 1986.
- 113. Heaton RK, Marcotte TD, Mindt MR, Sadek J, Moore DJ, Bentley H, McCutchan JA, Reicks C, Grant I, Group H. The impact of HIV-associated neuropsychological impairment on everyday functioning. Journal of the International Neuropsychological Society: JINS. 2004;10(3):317-31. doi: 10.1017/S1355617704102130. PubMed PMID: 15147590.

- 114. Tuluc F, Meshki J, Spitsin S, Douglas SD. HIV infection of macrophages is enhanced in the presence of increased expression of CD163 induced by substance P. Journal of leukocyte biology. 2014. doi: 10.1189/jlb.4AB0813-434RR. PubMed PMID: 24577568.
- 115. Yi Y, Shaheen F, Collman RG. Preferential use of CXCR4 by R5X4 human immunodeficiency virus type 1 isolates for infection of primary lymphocytes. J Virol. 2005;79(3):1480-6. Epub 2005/01/15. doi: 79/3/1480 [pii]
- 10.1128/JVI.79.3.1480-1486.2005. PubMed PMID: 15650174; PubMed Central PMCID: PMC544090.
- 116. Mexas AM, Graf EH, Pace MJ, Yu JJ, Papasavvas E, Azzoni L, Busch MP, Di Mascio M, Foulkes AS, Migueles SA, Montaner LJ, O'Doherty U. Concurrent measures of total and integrated HIV DNA monitor reservoirs and ongoing replication in eradication trials. Aids. 2012;26(18):2295-306. Epub 2012/09/28. doi: 10.1097/QAD.0b013e32835a5c2f. PubMed PMID: 23014521.
- 117. O'Doherty U, Swiggard WJ, Jeyakumar D, McGain D, Malim MH. A sensitive, quantitative assay for human immunodeficiency virus type 1 integration. J Virol. 2002;76(21):10942-50. PubMed PMID: 12368337; PubMed Central PMCID: PMC136638.
- 118. Yu JJ, Wu TL, Liszewski MK, Dai J, Swiggard WJ, Baytop C, Frank I, Levine BL, Yang W, Theodosopoulos T, O'Doherty U. A more precise HIV integration assay designed to detect small differences finds lower levels of integrated DNA in HAART treated patients. Virology. 2008;379(1):78-86. doi: 10.1016/j.virol.2008.05.030. PubMed PMID: 18649912; PubMed Central PMCID: PMC2610678.
- 119. Graf EH, Mexas AM, Yu JJ, Shaheen F, Liszewski MK, Di Mascio M, Migueles SA, Connors M, O'Doherty U. Elite suppressors harbor low levels of integrated HIV DNA and high levels of 2-LTR circular HIV DNA compared to HIV+ patients on and off HAART. PLoS pathogens. 2011;7(2):e1001300. doi: 10.1371/journal.ppat.1001300. PubMed PMID: 21383972; PubMed Central PMCID: PMC3044690.
- 120. Liszewski MK, Yu JJ, O'Doherty U. Detecting HIV-1 integration by repetitive-sampling Alu-gag PCR. Methods. 2009;47(4):254-60. doi: 10.1016/j.ymeth.2009.01.002. PubMed PMID: 19195495; PubMed Central PMCID: PMC2862469.
- 121. Eriksson S, Graf EH, Dahl V, Strain MC, Yukl SA, Lysenko ES, Bosch RJ, Lai J, Chioma S, Emad F, Abdel-Mohsen M, Hoh R, Hecht F, Hunt P, Somsouk M, Wong J, Johnston R, Siliciano RF, Richman DD, O'Doherty U, Palmer S, Deeks SG, Siliciano JD. Comparative analysis of measures of viral reservoirs in HIV-1 eradication studies. PLoS pathogens. 2013;9(2):e1003174. doi: 10.1371/journal.ppat.1003174. PubMed PMID: 23459007: PubMed Central PMCID: PMC3573107.
- 122. Hedeker D, Mermelstein RJ, Weeks KA. The thresholds of change model: an approach to analyzing stages of change data. Annals of behavioral medicine: a publication of the Society of Behavioral Medicine. 1999;21(1):61-70. doi: 10.1007/BF02895035. PubMed PMID: 18425656.
- 123. Vasan S, Poles MA, Horowitz A, Siladji EE, Markowitz M, Tsuji M. Function of NKT cells, potential anti-HIV effector cells, are improved by beginning HAART during acute HIV-1 infection. International immunology. 2007;19(8):943-51. doi: 10.1093/intimm/dxm055. PubMed PMID: 17702988.
- 124. Alter G, Malenfant JM, Delabre RM, Burgett NC, Yu XG, Lichterfeld M, Zaunders J, Altfeld M. Increased natural killer cell activity in viremic HIV-1 infection. Journal of immunology. 2004;173(8):5305-11. PubMed PMID: 15470077.
- 125. Della Chiesa M, Marcenaro E, Sivori S, Carlomagno S, Pesce S, Moretta A. Human NK cell response to pathogens. Seminars in immunology. 2014;26(2):152-60. doi: 10.1016/j.smim.2014.02.001. PubMed PMID: 24582551.
- 126. Bisio F, Bozzano F, Marras F, Di Biagio A, Moretta L, De Maria A. Successfully treated HIV-infected patients have differential expression of NK cell receptors (NKp46 and NKp30) according to AIDS status at presentation. Immunology letters. 2013;152(1):16-24. doi: 10.1016/j.imlet.2013.03.003. PubMed PMID: 23538009.
- 127. Finney CA, Ayi K, Wasmuth JD, Sheth PM, Kaul R, Loutfy MR, Kain KC, Serghides L. HIV infection deregulates innate immunity to malaria despite combination antiretroviral therapy. AIDS. 2013;27(3):325-35. doi: 10.1097/QAD.0b013e32835b3dfa. PubMed PMID: 23291537.
- 128. Deeks SG, Lewin SR, Havlir DV. The end of AIDS: HIV infection as a chronic disease. Lancet. 2013;382(9903):1525-33. Epub 2013/10/25. doi: S0140-6736(13)61809-7 [pii] 10.1016/S0140-6736(13)61809-7. PubMed PMID: 24152939.
- 129. Lopresti AL, Maker GL, Hood SD, Drummond PD. A review of peripheral biomarkers in major depression: the potential of inflammatory and oxidative stress biomarkers. Progress in neuro-psychopharmacology & biological psychiatry. 2014;48:102-11. doi: 10.1016/j.pnpbp.2013.09.017. PubMed PMID: 24104186.
- 130. Hunt PW. HIV and inflammation: mechanisms and consequences. Current HIV/AIDS reports. 2012;9(2):139-47. doi: 10.1007/s11904-012-0118-8. PubMed PMID: 22528766.

- 131. Tebas P, Tuluc F, Barrett JS, Wagner W, Kim D, Zhao H, Gonin R, Korelitz J, Douglas SD. A randomized, placebo controlled, double masked phase IB study evaluating the safety and antiviral activity of aprepitant, a neurokinin-1 receptor antagonist in HIV-1 infected adults. PLoS One. 2011;6(9):e24180. Epub 2011/09/21. doi: 10.1371/journal.pone.0024180
- PONE-D-11-07867 [pii]. PubMed PMID: 21931661; PubMed Central PMCID: PMC3169584.
- 132. Sperner-Unterweger B, Kohl C, Fuchs D. Immune changes and neurotransmitters: possible interactions in depression? Progress in neuro-psychopharmacology & biological psychiatry. 2014;48:268-76. doi: 10.1016/j.pnpbp.2012.10.006. PubMed PMID: 23085509.
- 133. Lichtblau N, Schmidt FM, Schumann R, Kirkby KC, Himmerich H. Cytokines as biomarkers in depressive disorder: current standing and prospects. International review of psychiatry. 2013;25(5):592-603. doi: 10.3109/09540261.2013.813442. PubMed PMID: 24151804.
- 134. Roff SR, Noon-Song EN, Yamamoto JK. The Significance of Interferon-gamma in HIV-1 Pathogenesis, Therapy, and Prophylaxis. Frontiers in immunology. 2014;4:498. doi: 10.3389/fimmu.2013.00498. PubMed PMID: 24454311; PubMed Central PMCID: PMC3888948.
- 135. Mackinnon DP, Lockwood CM, Williams J. Confidence Limits for the Indirect Effect: Distribution of the Product and Resampling Methods. Multivariate behavioral research. 2004;39(1):99. doi:
- 10.1207/s15327906mbr3901 4. PubMed PMID: 20157642; PubMed Central PMCID: PMC2821115.
- 136. MacKinnon DP. Introduction to statistical mediation analysis. New York: Lawrence Erlbaum Associates; 2008. x, 477 p. p.
- 137. Poli A, Michel T, Theresine M, Andres E, Hentges F, Zimmer J. CD56bright natural killer (NK) cells: an important NK cell subset. Immunology. 2009;126(4):458-65. doi: 10.1111/j.1365-2567.2008.03027.x. PubMed PMID: 19278419; PubMed Central PMCID: PMC2673358.
- 138. Said EA, Dupuy FP, Trautmann L, Zhang Y, Shi Y, El-Far M, Hill BJ, Noto A, Ancuta P, Peretz Y, Fonseca SG, Van Grevenynghe J, Boulassel MR, Bruneau J, Shoukry NH, Routy JP, Douek DC, Haddad EK, Sekaly RP. Programmed death-1-induced interleukin-10 production by monocytes impairs CD4+ T cell activation during HIV infection. Nature medicine.16(4):452-9. PubMed PMID: 20208540.
- 139. Uher R, Tansey KE, Dew T, Maier W, Mors O, Hauser J, Dernovsek MZ, Henigsberg N, Souery D, Farmer A, McGuffin P. An Inflammatory Biomarker as a Differential Predictor of Outcome of Depression Treatment With Escitalopram and Nortriptyline. The American journal of psychiatry. 2014. doi: 10.1176/appi.ajp.2014.14010094. PubMed PMID: 25017001.
- 140. Eller T, Vasar V, Shlik J, Maron E. Pro-inflammatory cytokines and treatment response to escitalopram in major depressive disorder. Progress in neuro-psychopharmacology & biological psychiatry. 2008;32(2):445-50. doi: 10.1016/j.pnpbp.2007.09.015. PubMed PMID: 17976882.
- 141. Lanquillon S, Krieg JC, Bening-Abu-Shach U, Vedder H. Cytokine production and treatment response in major depressive disorder. Neuropsychopharmacology. 2000;22(4):370-9. doi: 10.1016/S0893-133X(99)00134-7. PubMed PMID: 10700656.
- 142. Kraemer HC, Stice E, Kazdin A, Offord D, Kupfer D. How do risk factors work together? Mediators, moderators, and independent, overlapping, and proxy risk factors. The American journal of psychiatry. 2001;158(6):848-56. PubMed PMID: 11384888.
- 143. Molenberghs G, Verbeke G. Models for discrete longitudinal data. New York ; London: Springer; 2005. xxii, 683 p. p.
- 144. Nagelkerke N, Fidler V, Bernsen R, Borgdorff M. Estimating treatment effects in randomized clinical trials in the presence of non-compliance. Statistics in medicine. 2000;19(14):1849-64. PubMed PMID: 10867675.
- 145. Small DS, Ten Have TR, Joffe MM, Cheng J. Random effects logistic models for analysing efficacy of a longitudinal randomized treatment with non-adherence. Statistics in medicine. 2006;25(12):1981-2007. doi: 10.1002/sim.2313. PubMed PMID: 16220487.